CLINICAL TRIAL: NCT06549881
Title: Emergency Laparoscopic Cholecystectomy Guided by Indocyanine Green (ICG) Fluorescence: a Single Center Experience
Brief Title: Emergent Laparoscopic Cholecystectomy With ICG Cholangiography
Acronym: ELG-ICGC
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiaofei Liu, Clinical Associate professor, Peking Union Medical College Hospital
Other Study IDs: K5730-K24C2175
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Acute Cholestatic Hepatitis
Keywords: Emergent laparscopic cholecystectomy; indocyanine green fluorescence; surgical outcome; economic effectiveness; acute cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICG fluorescence guided group: Patients with acute cholecystitis underwent emergent laparscopic cholecystectomy guided by indocyanine green (ICG) fluorescence.
  Interventions: Procedure: emergency laparoscopic cholecystectomy guided by indocyanine green (ICG) fluorescence

INTERVENTIONS:
Procedure: emergency laparoscopic cholecystectomy guided by indocyanine green (ICG) fluorescence — emergency laparoscopic cholecystectomy guided by indocyanine green (ICG) fluorescence

SUMMARY:
A consecutive case series report to share our experience in surgical outcome of patients who underwent emergency laparoscopic cholecystectomy guided by indocyanine green (ICG) fluorescence. The patients were recruited in PUMCH emergency department from 2023 to 2024.

DETAILED DESCRIPTION:
Acute calculous cholecystitis, typically occurs in patients with gallstones, accounts for 90 to 95% of acute cholecystitis. Emergent laparscopic cholecystectomy (ELC) is the major treatment option. Traditionally, the time frame for ELC is generally considered to be within 72 hours from the onset of symptoms. However, with the development of surgical techniques, nowadays, ELC is also considered for patients with symptoms onset within 10 days and hospital stays within 7 days. The determination of the time frame for ELC in acute cholecystitis is primarily based on the risk of complications occurring. Comparing to delayed laparscopic cholecystectomy (DLC), ELC has advantages in post-operative complications in patients with symptoms onset within 72 hours. Post-operative complications for both DLC and ELC include bile leaks, intestinal obstruction, ascites, intraperitoneal hemorrhage, would bleeding and hematoma, wound infection and calculus remaining. Most of them associate with intraoperative procedures. Laparoscopic cholecystectomy guided by indocyanine green (ICG) fluorescence, comparing to conventional laparscopic procedures, can help the surgeons to identify bile tracts and therefore may reduce the complications. Therefore, we conduct this case series report to share our single center experience of surgical outcomes and economic effectiveness of laparoscopic cholecystectomy guided by ICG.

The surgical outcomes are evaluated by both intraoperative events and postoperative events. Intraoperative events contain the following items: (1) incidence of intraoperative accidental bile tract injury, (2) intraoperative bleeding (volume), (3) operation time. Postoperative events contain the following items: (1) incidence of complications staging 2 and above according to Clavien Dindo Grade during hospital stay, (2) duration of postoperative hospital stay. The economic effectiveness is evaluated by cost of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All of the hospitalized patients of underwent emergent laparscopic cholecystectomy guided by ICG fluorescence by the emergent surgeon team from 1st August 2023 to 1st Feburary 2024 in the department of Emergency in Peking Union Medical College Hospital

Exclusion Criteria:

* Patients with incomplete medical records. Patients have other emergent conditions which warrant other emergent operations or major treatment simultaneously besides ELC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute cholecystitis warrant emergent laparscopic cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
incidence of intraoperative accidental bile tract injury | within 1 month after after discharge
  The primary outcome is incidence of intraoperative accidental injury involving the bile tract in emergent laparscopic cholecystectomy guided by ICG fluorescence. The injury manifests as biliary obstruction, biliary leak, or biliary stricture. Medical records will be reviewed to identify an intraoperative bile tract injury event.
incidence of postoperative complications | within 1 month after discharge
  incidence of complications staging 2 and above according to Clavien Dindo Grade during hospital stay

SECONDARY OUTCOMES:
duration of postoperative hospital stay | within 1 month after discharge
  Days of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Qiaofei Liu, M.D, Principal Investigator — Department of General Surgery, Peking Union Medical College Hospital
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No